CLINICAL TRIAL: NCT00344604
Title: The Role of Psychosocial and Other Quality of Life Parameters in Evaluating Functional Changes Prior to and Following Laser In-situ Keratomileusis (LASIK)
Brief Title: The Role of Psychosocial and Other Quality of Life Parameters in Evaluating Functional Changes Prior to and Following Laser In-situ Keratomileusis (LASIK)Changes Laser In-situ Keratomileusis (LASIK)
Status: Withdrawn | Type: Observational
Why Stopped: PI decided to terminate the study at this time
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: James P. McCulley, UTSW Medical Center at Dallas
Other Study IDs: 032004-028
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Keratomileusis, Laser In Situ
Keywords: Patients who have undergone routine LASIK as a primary refractive procedure for myopia, hyperopia, or astigmatism.
MeSH Terms: conditions — Hyperopia; Astigmatism

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Role of psychosocial and quality of life parameters prior to and following LASIK.

SUMMARY:
To evaluate the changes in quality of life parameters after LASIK surgery.

DETAILED DESCRIPTION:
Our purpose is to evaluate the changes in quality of life parameters after LASIK surgery. We intend to create a questionnaire to delineate the changes that occur in LASIK patients at the pre-operative visit and at the 1-month and 3-month post-operative visits. Additional questionnaires will be administered to demonstrate the validity of the new questionnaire. The approximate time the patient will be required to spend in clinic will be approximately 45 minutes at each of the three visits.

ELIGIBILITY:
Inclusion Criteria: All refractive surgery patients with otherwise normal eyes undergoing routine LASIK as a primary refractive procedure for myopia, hyperopia or astigmatism.

-

Exclusion Criteria: Patients who elect to perform alternative refractive surgery such as PRK, RK, or Intacts™.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-03; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shady Awwad, M.D., Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States